CLINICAL TRIAL: NCT02825849
Title: Platelet-rich Plasma (PRP) for Endometrial Regeneration and Repair: a Prospective Randomised Pilot Study
Brief Title: Platelet-rich Plasma (PRP) for Endometrial Regeneration and Repair
Acronym: PRP-E
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment and competing studies have published.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-19764
Record Dates: First submitted 2016-07-03; First posted 2016-07-07 (Estimated); Results first posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Infertility; Asherman's Syndrome
Keywords: endometrium; thin uterine lining; uterine scarring
MeSH Terms: conditions — Infertility; Gynatresia

STUDY DESIGN:
Intervention Model Description: During Study Period #1: Subjects were randomized to receive either PRP or standard care. A total of 13 subjects were randomized.
  The study design was then altered to remove randomization (10/4/2018). All patients in Study Period #2 received PRP. An additional 14 subjects were enrolled in Study Period #2.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRP intrauterine infusion (Experimental): Intrauterine infusion of platelet rich plasma in combination with standard treatment, in patients with Asherman's Syndrome or thin uterine lining in frozen embryo transfer cycles
  Interventions: Biological: Intrauterine infusion of platelet rich plasma
- Control group with standard treatment only (No Intervention): Patients with Asherman's Syndrome or thin uterine lining in frozen embryo transfer cycles undergoing standard treatment protocols

INTERVENTIONS:
Biological: Intrauterine infusion of platelet rich plasma — Patients randomized to study group will have 30cc of blood drawn with isolation of platelet rich plasma (PRP) per standard manufacturer's protocol, with subsequent intrauterine infusion of this autologous PRP.
  Other Names: PRP
  Arms: PRP intrauterine infusion

SUMMARY:
Patients with intrauterine adhesions (Asherman's Syndrome) and persistent thin endometrial lining in in vitro fertilization (IVF) treatment programs, particularly those resistant to standard therapies, present a significant clinical challenge. The aim of this trial is to assess if intrauterine administration of platelet rich plasma (PRP) improves endometrial lining thickness in patients with thin lining or Asherman's Syndrome.

DETAILED DESCRIPTION:
BACKGROUND:

There is a need for new and more effective therapies for patients with intrauterine adhesions (Asherman's Syndrome) and persistent thin endometrial lining in in vitro fertilization (IVF) treatment programs, particularly for patients resistant to standard therapies

HYPOTHESIS:

Platelet rich plasma stimulates cellular processes involved in endometrial regeneration relevant to management of a thin lining or intrauterine scarring.

PRIMARY AIMS:

- To measure the change in endometrial lining thickness

SECONDARY AIMS:

* To determine if fertility is improved in patients receiving platelet rich plasma (PRP):

  1. In patients with thin lining undergoing frozen embryo transfer (FET), to determine:
* clinical pregnancy rate

  2. In patients with Asherman's Syndrome, to determine:
* the chance of spontaneous pregnancy

Any adverse effects of study arm will be monitored and reported as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Persistent thin lining < 6mm on >1 cycle in previous IVF or FET cycle OR moderate-to-severe Asherman's syndrome

Exclusion Criteria:

* Age <18 years old or >43 years old,
* Pregnancy,
* Diagnosis of cancer,
* Hb <11 g/dL, platelets <150,000/mm3,
* Anticoagulation,
* NSAIDs in the 10 days before procedure
* Any significant comorbidity or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
* Incision in the uterus: myomectomy; cesarean section

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-11; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather G. Huddleston, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco - Center for Reproductive Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PRP Intrauterine Infusion | Control Group With Standard Treatment Only
Started | 22 | 5
Completed | 22 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRP Intrauterine Infusion | Control Group With Standard Treatment Only | Total
Number analyzed (Participants) | 22 | 5 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (3.2) | 35.6 (6.3) | 37.5 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 5 | 27
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 5 | 27
Endometrial Thickness [Mean (Standard Deviation); unit: cm] | 6.3 (2.3) | 4.3 (1.2) | 5.9 (2.3)
Ashermans score on hysteroscopy [Mean (Standard Deviation); unit: score] — The American Fertility Society (presently ASRM) developed a classification system upon hysteroscopic assessment of intrauterine adhesions. Parameters assessed are: extent of cavity involved (<1/3, 1/3-2/3 an >2/3, with scores 1, 2, 4 respectively), type of adhesions (filmy, filmy and dense and dense, with scores 1, 2, 4 respectively), menstrual pattern (normal, hypomenorrhea, amenorrhea, with scores 0, 2, 4 respectively). Then overall severity of intrauterine adhesive disease is expressed as a total: stage 1 (mild) - score 1-4, Stage II (moderate (score 5-8), Stage III (severe)- score 9-12. Population: This score was only calculated for patients with ashermans syndrome who had hysteroscopy in the randomized trial portion of the study.
  score
    number analyzed (Participants) | 8 | 5 | 13
    (all) | 5.6 (1.17) | 5.8 (2.49) | 5.67 (1.63)

OUTCOME MEASURES:

1. Primary Outcome: Endometrial Thickness
Description: Endometrial thickness will be measured using transvaginal ultrasound per standard protocol
Time Frame: 3-30 days after treatment
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | PRP Intrauterine Infusion | Control Group With Standard Treatment Only
Number analyzed (Participants) | 22 | 5
cm | 6.4 (2.4) | 5.2 (2.3)

2. Secondary Outcome: Number of Participants With Ultrasound Confirmed Clinical Pregnancies
Description: Defined by ultrasound confirmed pregnancies per total participants in each arm
Time Frame: at least 7 weeks after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | PRP Intrauterine Infusion | Control Group With Standard Treatment Only
Number analyzed (Participants) | 22 | 5
Participants | 12 | 3
Statistical Analysis 1: Comparison: PRP Intrauterine Infusion vs Control Group With Standard Treatment Only; Test type: Superiority; p = .824, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events were collected for up to 365 days after study treatment
Arm/Group | PRP Intrauterine Infusion | Control Group With Standard Treatment Only
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/5
Other Adverse Events (participants affected / at risk) | 0/22 | 0/5

LIMITATIONS AND CAVEATS:
The study was a pilot study and was not adequately powered to detect a difference. In addition the study was closed prior to full enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2020-11-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT02825849/SAP_000.pdf
  • Study Protocol (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT02825849/Prot_001.pdf
  • Informed Consent Form (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT02825849/ICF_002.pdf